CLINICAL TRIAL: NCT01904461
Title: Monocentric, Prospective, Comparative and Randomised Study on the Use of a Haemostatic Vacuum Device During Tonsillectomy in Children
Brief Title: HemORL: Monocentric, Prospective, Comparative Study on the Use of a Haemostatic Vacuum Device During Tonsillectomy in Children
Acronym: HemORL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: HEMOSQUID (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HemORL-DCIC-1211
Record Dates: First submitted 2013-07-05; First posted 2013-07-22 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Tonsillectomy; Hemorrhage; Postoperative Complications
Keywords: tonsillectomy; children; vacuum; medical device; pain; hemorrhage; post-surgical complications
MeSH Terms: conditions — Hemorrhage; Postoperative Complications; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vacuum device surgery (Experimental): At first the surgeon proceed to the dissection of children tonsils and at last he uses the innovative vacuum device to obtain wounds hemostasis
  Interventions: Device: Vacuum device
- Conventional surgery (Active Comparator): At first the surgeon proceed to the dissection of children tonsils and at last he uses a bipolar forceps to obtain wounds hemostasis
  Interventions: Procedure: Conventional surgery

INTERVENTIONS:
Device: Vacuum device
  Other Names: -Suction cup; -Redon 600ml
  Arms: Vacuum device surgery
Procedure: Conventional surgery
  Arms: Conventional surgery

SUMMARY:
The long-term objective of this study is to prove:

* the equivalence of the number of post-operation hemorrhages, and maybe a decrease of the number of secondary hemorrhages
* the decrease of pain and quicker re-feeding
* an easier haemostasis
* the simplification of the tonsillectomy surgical kit
* the decrease of dissection time

ELIGIBILITY:
Inclusion Criteria:

* children from 3 to 10 years old undergoing tonsillectomy (with or without adenoidectomy)
* children without known hemophilia or any coagulation trouble
* children speaking and understanding French
* children's both parents must speak and understand French
* children's both parents must be affiliate to social security or similarly regime

Exclusion Criteria:

* children with known allergy to silicone
* refusal to consent: from child's age to consent or from both parents
* telephone monitoring refusal
* protected person referred to in Articles L1121-6 of the Code of Public Health
* children's both parents are protected persons referred to in Articles L1121-8 of the Code of Public Health

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-09 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of cauterization time to obtain the tonsillectomy wounds hemostasis using bipolar forceps between conventional surgery group and the vacuum device group | From the beginning to the end of a tonsillectomy: an expected average of 2 hours
  Cauterization time (seconds) needed to obtain wounds tonsillectomy hemostasis using bipolar forceps(electric power of 20W)

SECONDARY OUTCOMES:
Assessment of the vacuum device hemostatic technique at his installation on the wound | From the beginning to the end of a tonsillectomy: an expected average of 2 hours
  * Number of success or failure to install the device
  * Cases of no immediately hemostasis
Assessment between two arm of the postoperative pain until 10 days after the surgery | 10 days
  Pain score every day (FLACC -> children between 3 and 7 years old Faces pain scale -> children between 8 and 10 years old)
Comparison of the time of the first complaint of pain after surgery between conventional surgery group and the vacuum device group | Time between general anesthesia and discharge hospitalization: an average of one day
  Time between general anesthesia and first complaint of pain
Comparison of surgery time between the 2 arm | An expected average of 2 hours
  Time between the first incision and final wounds hemostasis verification
Comparison between the 2 arms of re-feeding without pain (liquids,semi-liquids ands solids) | Until 11 days after surgery
  Time or/and day of the first meal without pain
Comparison between the 2 arms of the number of primary hemorrhages | Until 24 hours after surgery
  Number of primary hemorrhages
Comparison between the 2 arms of the number of secondary hemorrhages | From 24 hours after surgery until 11 days after surgery
  Number of secondary hemorrhages
Comparison between the 2 arms of the number of rehospitalisation (all circumstances) | From 24 hours after surgery until 11 days after surgery
  Number of rehospitalisation
Comparison between the 2 arms of the number of strong analgesics doses | Until 11 days after surgery
  Number of strong analgesics doses per day. Strong analgesics are used only if the child has a FLACC score higher than 3 (children from 3 to 7 years old) and a Faces Pain Scale score higher than 4 (children from 8 to 10 years old).
Clinician evaluation about the feasibility of the vacuum device installation | From the beginning to the end of a tonsillectomy: an expected average of 2 hours
  Score from a qualitative satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Schmerber, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, Grenoble, Isère, France

REFERENCES:
- [Background] Guerrero K, Moreau-Gaudry A, Porcu P, Blin D. An innovative technique to control bleeding with vacuum device. Eur J Cardiothorac Surg. 2011 Jun;39(6):1070-2. doi: 10.1016/j.ejcts.2010.09.047. Epub 2010 Nov 12. PMID 21075003
- [Background] Brichon PY, Porcu P, Moreau-Gaudry A, Blin D. Extraction of substernal goitre using an innovative vacuum device. Eur J Cardiothorac Surg. 2012 Jul;42(1):178-9. doi: 10.1093/ejcts/ezs018. Epub 2012 Feb 13. PMID 22334630
- [Background] Porcu P, Moreau-Gaudry A, Chavanon O, Blin D. Haemostasis of a right ventricle-gunshot wound using a novel haemostatic vacuum device. Interact Cardiovasc Thorac Surg. 2012 Aug;15(2):294-6. doi: 10.1093/icvts/ivs103. Epub 2012 May 7. PMID 22566511
- See also: Website of the Grenoble clinical investigation center - Technological Innovation — http://www.cic-it-grenoble.fr/